CLINICAL TRIAL: NCT02878499
Title: Do Sleep and Circadian Rhythm Disturbances Impact the Cognitive and Behavioural Development of Children With Autism?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5060
Record Dates: First submitted 2016-06-14; First posted 2016-08-25 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; autism spectrum disorder; ASD; sleep; Circadian; Biological rhythms; melatonin; Cognition; Behavior; Longitudinal; Longitudinal accelerated design
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASD (Other)
  Interventions: Other: polysomnography

INTERVENTIONS:
Other: polysomnography

SUMMARY:
The primary objective of this study is to undertake a longitudinal investigation of the impact of sleep and circadian rhythm disturbances on cognitive and behavioural trajectories in children with autism spectrum disorder (ASD) age 3-10 years old.

This innovative study will use objective quantifiable measures of sleep and circadian rhythms in addition to subjective measures.

The investigators aim to assess the hypotheses that, in pre-pubertal children with ASD,

1. sleep disturbances are correlated with circadian rhythm disturbances;
2. both sleep and circadian rhythm disturbances are negatively correlated with cognitive performance and positively correlated with behavioural disturbances;
3. sleep and circadian rhythm disturbances, most notably abnormal melatonin secretion, impact the cognitive and behavioural development of children with ASD, depending on age (prospective longitudinal analyses).

ELIGIBILITY:
Inclusion criteria:

* Age: from 3 to 8 years of age at inclusion, as per defined entry ages (longitudinal accelerated design)
* Diagnostic criteria of autism spectrum disorder (ASD)
* Autism Diagnostic Interview (ADI) - revised (R) score compatible with ASD diagnosis
* Autism Diagnostic Observation Schedule (ADOS) score compatible with ASD diagnosis
* Study information has been understood
* Study consent signed by both parents or legal representatives and by the child if the child is capable of expressing his consent
* Stable medication over the 2 months-period preceding inclusion and during evaluation periods (exception: (1) medication mentioned in the exclusion criteria, (2) a new medication instaurated between two evaluation periods is not in itself an exclusion criteria, but will be taken into account in data analysis)
* Compliance with study procedures
* Priori clinical medical examination
* Child affiliated with social security Concerning sleep disorders: the discovery of a primary sleep disorder (e.g.: sleep apnea syndrome, restless legs syndrome, periodic limb movements during sleep) as well as their treatment is not a criteria for terminating the study but will be taken into account in data analysis

Exclusion criteria:

* Secondary autism: e.g. associated with Rett syndrome, fragile X syndrome, Down syndrome, Bourneville tuberous sclerosis, von Recklinghausen disorder, Cytomegalovirus (CMV) encephalitis, congenital rubeola, phenylketonuria.
* Current treatment with melatonin or melatonin agonists before study entry (before baseline assessment)
* Changes in medication over the 2 months-period preceding the study (exception: a new medication instaurated between two evaluation periods is not in itself an exclusion criteria, but will be taken into account in data analysis)
* Transmeridian travel (> 2 time zones) in the month preceding the study
* Participation in other research studies in the 3 months period preceding the study
* Treatment with betablockers, local or systemic non-steroidal anti-inflammatory (NSAI) agents, benzodiazepines, antidepressants
* Severe other intercurrent disorder.
* Severe allergies.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2012-12-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in sleep latency at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Sleep latency derived from actigraphy
Change in sleep fragmentation index at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Sleep fragmentation index derived from polysomnography (PSG)
Change in nocturnal melatonin secretion at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Nocturnal melatonin secretion (6-SMT measured in night urine from 8pm to 8am)
Change in amplitude of the day-night melatonin secretion at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Amplitude of the day-night melatonin secretion (6 sulfatoxy-melatonin (6-SMT) measured in 12h-night versus 12h-day urine)
Change in non-verbal index (INV, derived from the Kaufmann-Assessment Battery fir Children II (K-ABC II)) at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Change in verbal intelligence quotient (IQ) at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Change in verbal intelligence quotient (IQ) derived from the appropriate Wechsler scales for children (WPPSI or WISC) at 1 year follow-up and 2 year follow-up compared to baseline
Change in Raven performance IQ at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Raven performance IQ derived from Raven progressive matrices (CPM-BF) at 1 year follow-up and 2 year follow-up compared to baseline
Change in Autism Diagnostic Observation Schedule (ADOS), module 1-3: part 'D' et 'E' (repetitive and abnormal behaviour) at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Change in aberrant Behaviour Checklist (ABCL) global score at 1 year follow-up and 2 year follow-up compared to baseline | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up

SECONDARY OUTCOMES:
presence of an intrinsic sleep disorders (e.g. obstructive or central sleep apnea syndrome, restless legs syndrome and periodic limb movements during sleep…) | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Total sleep time (TST) | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Time and percentage of TST spent in different sleep stages (slow wave sleep, rapid eye movement (REM) sleep) | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Sleep spindle density in light slow wave sleep | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Density of rapid eye movements in REM sleep | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Spectral analysis of the sleep electro-encephalogram (EEG) | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
24h urinary 6-sulfatoxymelatonin levels (ng/ml) | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Inter-daily stability (IS) and intra-daily variability (IV) of circadian rhythms (actigraphy derived) | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
  Level of ferritin in plasma
Circadian phase of body temperature | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up
Level of ferritin in plasma | Three annual assessments: baseline, 1 year follow-up, 2 year follow-up

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Lyon - CHS Le Vinatier, Lyon
  - CHU Gui de Chaulhiac, Montpellier
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de TOURS - Hôpital Bretonneau, Tours